CLINICAL TRIAL: NCT00872222
Title: Uncontrolled Prospective Multi-Centre Post Marketing Surveillance Study to Monitor the Long Term Survivorship of Pinnacle™ Acetabular Cup Prosthesis With a Ceramic-on-ceramic Bearing in Subjects With Aetiologies Requiring a Primary Total Hip Replacement
Brief Title: A Single Centre Study to Assess the Long-term Performance of the Pinnacle™ Cup With a Ceramic-on-ceramic Bearing in Primary Total Hip Replacement
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study terminated early due to business reasons
Sponsor: DePuy International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT03/39
Record Dates: First submitted 2009-03-30; First posted 2009-03-31 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-09

CONDITIONS: Rheumatoid Arthritis; Osteoarthritis; Post-traumatic Arthritis; Collagen Disorders; Avascular Necrosis; Traumatic Femoral Fractures; Nonunion of Femoral Fractures; Congenital Hip Dysplasia; Slipped Capital Femoral Epiphysis
Keywords: Hip; Cementless; Ceramic-on-Ceramic
MeSH Terms: conditions — Arthritis, Rheumatoid; Osteoarthritis; Collagen Diseases; Osteonecrosis; Hip Dislocation, Congenital; Slipped Capital Femoral Epiphyses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ceramic-on-Ceramic (Other): Pinnacle™ Acetabular System with ceramic liner
  Interventions: Device: Pinnacle™ Acetabular System

INTERVENTIONS:
Device: Pinnacle™ Acetabular System — A cementless acetabular cup with ceramic liner for use in total hip replacement

SUMMARY:
The purpose of this study is to monitor the performance of the Pinnacle™ Cup with a ceramic-on-ceramic bearing combination in the treatment of patients with hip joint disease requiring a total hip replacement. Patients who enter the study will be evaluated at regular intervals following hip surgery using patient, clinical and x-ray assessments.

ELIGIBILITY:
Inclusion Criteria:

i) Male or female subjects, aged between 18 and 70 years inclusive.

ii) Subjects who are able to give voluntary, written informed consent to participate in this investigation and from whom consent has been obtained.

iii) Subjects who, in the opinion of the Investigator, are able to understand this investigation, co-operate with the investigational procedures and are willing to return to the hospital for all the required post-operative follow-ups.

iv) Subjects undergoing primary total hip replacement who are suitable for cementless acetabular components.

Exclusion Criteria:

i) Subjects who, in the opinion of the Investigator, have an existing condition that would compromise their participation and follow-up in this study.

ii) Subjects undergoing revision hip replacement.

iii) Women who are pregnant.

iv) Subjects who are known drug or alcohol abusers or with psychological disorders that could effect follow-up care or treatment outcomes.

v) Subjects who have participated in a clinical study with an investigational product in the last 12 months.

vi) Subjects who are currently involved in any injury litigation claims.

vii) Subjects undergoing a simultaneous bilateral hip operation.

viii) Subjects undergoing the second stage of a staged bilateral for whom the contralateral hip is part of this clinical investigation.

ix) Subjects undergoing the second stage of a staged bilateral for whom the contralateral hip was implanted less than six months previously or is not performing satisfactorily

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2007-01; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Kaplan-Meier survivorship at the five-year period | 5yrs

SECONDARY OUTCOMES:
Kaplan-Meier survivorship calculations | Annually
Harris Hip Score | 6mths, 1yr, 2yrs, 5yrs, 7yrs, 10yrs and 15yrs post-surgery
Radiographic analysis | 6mths, 1yr, 2yrs, 5yrs, 7yrs, 10yrs and 15yrs post-surgery
Oxford Hip score | 3yrs, 4yrs, 6yrs, 8yrs, 9yrs, 11yrs, 12yrs, 13yrs and 14yrs post-surgery

CONTACTS AND LOCATIONS:
Locations (1):
- St Anne's University Hospital, Brno, Czechia